CLINICAL TRIAL: NCT06121609
Title: The 90% Effective Dose (ED90) of Remimazolam Anesthesia Induction in Painless Bidirectional Endoscopy in Children: a Biased Coin up and Down Sequential Trial
Brief Title: ED90 of Remimazolam Anesthesia Induction in Painless Bidirectional Endoscopy in Children
Acronym: ED90
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Doctor, Tongji Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EDRC
Record Dates: First submitted 2023-10-25; First posted 2023-11-08 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Bidirectional Endoscopy
Keywords: pediatric anesthesia; remimazolam; ED90
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4-6 years group (Experimental): Age: ≥48 and <84 months
  Interventions: Drug: Remimazolam
- 7-12 years group (Experimental): Age: ≥84and <156 months
  Interventions: Drug: Remimazolam
- infant group (Experimental): Age: <48 months
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Exploring ED90 induced by remimazolam anesthesia in children of different age groups undergoing painless bidirectional endoscopy
  Other Names: Remimazolam besylate

SUMMARY:
Exploring the ED90 of remimazolam in pediatric bidirectional endoscopy at different age groups.

DETAILED DESCRIPTION:
Exploring the ED90 of remimazolam in pediatric bidirectional endoscopy at different age groups, providing a more scientific clinical dose selection basis for the anesthesia induction application of Remazolam.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-12 years old,
2. ASA I-II level;
3. Sign an informed consent form.

Exclusion Criteria:

1. Developmental delay or neurological and psychiatric disorders;
2. Severe malnutrition or severe obesity;
3. High risk of stomach fullness and reflux aspiration;
4. Allergic to benzodiazepines and opioids;
5. Those who have taken sedative, analgesic, or antidepressant drugs within 24 hours;
6. Severe sleep apnea;
7. Abnormal liver and kidney function;
8. Recently participated in other clinical studies.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: aihua Du, Dr., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
You can request it from the main researcher.

REFERENCES:
- [Derived] Zhou SQ, Bi Y, Chu TT, Tian Z, Yu SC, Yan TQ, Deng JB, Xu AJ. Effective remimazolam induction dose in paediatric same-day bidirectional endoscopy: A biased coin up and down sequential trial. Br J Clin Pharmacol. 2025 Dec 4. doi: 10.1002/bcp.70406. Online ahead of print. PMID 41342333

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4-6 Years Group | 7-12 Years Group | Infant Group
Started (The initial sample size is the sample size that this study expects to include in the sequential experimental order.) | 55 | 55 | 55
Completed | 55 | 55 | 10
Not Completed | 0 | 0 | 45
Not completed — Lack of Efficacy | 0 | 0 | 45

BASELINE CHARACTERISTICS:
Population: The infant group was terminated early due to unknown safety dose boundaries.
Groups:
- Total: Total of all reporting groups
Arm/Group | 4-6 Years Group | 7-12 Years Group | Infant Group | Total
Number analyzed (Participants) | 55 | 55 | 10 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 55 | 55 | 10 | 120
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6 [4.95 to 6] | 9 [8 to 11] | 3 [2.8 to 3.5] | 6 [5.95 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 3 | 48
  Male | 32 | 33 | 7 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 55 | 55 | 10 | 120
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 55 | 55 | 10 | 120
BMI [Mean (Standard Deviation); unit: kg/m2] | 15 (1.58) | 17 (2.49) | 15 (1.96) | 16 (2.12)

OUTCOME MEASURES:

1. Primary Outcome: Modified Observer's Assessment of Alertness/Sedation Scale, MOAA/S
Description: Using the modified MOAA/S scoring table（ranging from 5-0） to evaluate if the sedation is successful.
  5 points：Respond quickly to names spoken in a normal tone 4 points：Showing a drowsy reaction to names spoken in a normal tone 3 points：Only react after loudly and/or repeatedly calling the name 2 points：Response immediately after slight stimulation or shaking
  1point：Response only occurs after compression of the trapezius muscle that causes pain 0 point：No response after compression of the trapezius muscle
Time Frame: The entire duration of anesthesia：From the start of drug administration for induction until the patient's awakening.
Population: The infant group was terminated prematurely due to the unknown safety dose boundary.
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | 4-6 Years Group | 7-12 Years Group | Infant Group
Number analyzed (Participants) | 55 | 55 | 10
units on a scale | 0.674 [0.66 to 0.76] | 0.449 [0.423 to 0.59] | 0.937 [0.65 to 1.264]

2. Secondary Outcome: Respiratory Suppression Incidence
Description: Respiratory frequency<8 times/min or SP02<90%
Time Frame: The entire duration of anesthesia：From the start of drug administration for induction until the patient's awakening.
Measure: Count of Participants; unit: Participants
Arm/Group | 4-6 Years Group | 7-12 Years Group | Infant Group
Number analyzed (Participants) | 55 | 55 | 10
Participants | 4 | 7 | 2

3. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Intraoperative blood pressure and heart rate changes: record the patient's intraoperative blood pressure, heart rate, and the use of related vasoactive drugs; Postoperative adverse reactions: such as hypertension, hypotension, tachycardia, gastrointestinal symptoms, postoperative restlessness, etc.
Time Frame: From the start of drug administration for induction to 24h after the operation.
Measure: Count of Participants; unit: Participants
Arm/Group | 4-6 Years Group | 7-12 Years Group | Infant Group
Number analyzed (Participants) | 55 | 55 | 10
Participants | 0 | 0 | 0

4. Secondary Outcome: Time Records
Description: induction time
Time Frame: The entire duration of anesthesia：From the start of drug administration for induction until the patient's awakening.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | 4-6 Years Group | 7-12 Years Group | Infant Group
Number analyzed (Participants) | 55 | 55 | 10
seconds | 120 [80 to 140] | 100 [80 to 120] | 150 [125 to 175]

ADVERSE EVENTS:
Time Frame: 3days
Description: The infant group was terminated prematurely due to the unknown safety dose boundary.
Arm/Group | 4-6 Years Group | 7-12 Years Group | Infant Group
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/10
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT06121609/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT06121609/ICF_001.pdf